CLINICAL TRIAL: NCT02565069
Title: Identification for the Treatment of Complex Arrhythmias (CartoFinder™ Algorithm Trial: "CF163 EU")
Brief Title: Identification for the Treatment of Complex Arrhythmias
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIND-EU - CF163
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment group (Experimental): Use of CartoFinder™ device with CARTO® 3 System V5 Navigation to treat complex arrhythmias
  Interventions: Device: CartoFinder™ Device with CARTO® 3 System V5 Navigation

INTERVENTIONS:
Device: CartoFinder™ Device with CARTO® 3 System V5 Navigation — Ablation treatment

SUMMARY:
The primary purpose of this trial is to demonstrate that the utilization of CartoFinder™ 4D Local Activation Time (LAT) Algorithm may help identify and improve the outcome for the treatment of complex arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Signed the Patient Informed Consent Form (ICF)
3. Scheduled to undergo a clinically-indicated catheter ablation procedure for treatment of

   * Persistent atrial fibrillation (defined as continuous atrial fibrillation that is sustained beyond seven consecutive days).
   * Drug-resistant Atrial Fibrillation. (failed 1 or more class I or III antiarrhythmic drugs) and demonstrating Persistent AF (requiring drugs or electrical shock to terminate)
   * Persistent AF despite prior conventional ablation.
4. Previous procedure permitted but limited to single Pulmonary Vein Isolation (PVI).
5. In AF at the time of the Pre-CartoFinder Map (spontaneous or induced)
6. Able and willing to comply with all pre-, post-, and follow-up testing and requirements.

Exclusion Criteria:

1. Paroxysmal Atrial Fibrillation
2. Continuous AF > 12 months (1-Year) (Longstanding Persistent AF)
3. Cardioversion refractory (The inability to restore sinus rhythm for 30 secs or longer following electrical cardioversion. If a patient does not have documented evidence of being successfully cardioverted (Normal Sinus Rhythm (NSR) > 30 secs), the patient must be cardioverted prior to the ablation procedure. Failure to cardiovert based on the above criteria is considered a screen failure.
4. A complex arrhythmia secondary to a reversible or non-cardiac cause. For example: a complex arrhythmia secondary to electrolyte imbalance or thyroid disease.
5. Left atrial size >55 mm (echocardiography, parasternal long axis view).
6. Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study.
7. Structural atrial disease such as a prior history of atriotomy from prior atrial surgery, presence of an atrial septal defect, and/or presence of an atrial septal closure patch.
8. History of or current blood clotting or bleeding abnormalities, contraindication to systemic anticoagulation (i.e., heparin, warfarin, dabigatran, or a direct thrombin inhibitor), significant pulmonary disease, cardiac surgeries, unstable angina, uncontrolled heart failure, acute illness or systemic infection, or any other disease or malfunction that would preclude treatment in the opinion of the investigator.
9. Enrollment in an experimental study evaluating another device or drug under investigation.
10. Prosthetic valve
11. Presence of intramural thrombus, tumor or other abnormality / condition that precludes vascular access, catheter introduction or manipulation.
12. Women of child bearing potential whom are pregnant, lactating, or planning to become pregnant during the course of the trial.
13. Presenting contra-indications for the devices used in the study, as indicated in the respective Instructions For Use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-07-01; Primary Completion 2017-01-24 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
Identify rate of slowing for the overall mean atrial fibrillation rate | Day 0 (procedure date)
  Identify rate of slowing for the overall mean atrial fibrillation rate that can be achieved by using CARTOFINDER™ 4D LAT Algorithm
Evaluate Freedom from procedure-related primary adverse events | 7 days
  Evaluate Freedom from procedure-related primary adverse events at 7 days post-procedure

SECONDARY OUTCOMES:
Evaluate procedural results | Day 0 (procedure date)
  Proportion of subjects with focal impulses / Repetitive Activation Pattern (RAP)s and number of areas and locations of focal impulses / RAPs
Evaluate procedural results | Day 0 (procedure date)
  Proportion of subjects with Normal Sinus Rhythm (NSR) after CF guided ablation
Evaluate procedural results | Day 0 (procedure date)
  Proportion of subjects with AF organization after CF guided ablation
Evaluate procedural results | Day 0 (procedure date)
  Proportion of subjects with acute procedural success, i.e. subjects with spontaneous return to NSR or AF organization after CF guided ablation
Evaluate freedom from documented recurrence of atrial fibrillation | 6 and 12 months
  Evaluate freedom from documented recurrence of atrial fibrillation at 6 and 12 months post-procedure